CLINICAL TRIAL: NCT07095530
Title: Horizontal Ridge Augmentation Using Polyvinylidene Fluoride Versus Titanium Mesh Membranes - A Randomized Clinical Trial
Brief Title: Horizontal Ridge Augmentation Using Polyvinylidene Fluoride Versus Titanium Mesh Membranes
Acronym: PVDF + HRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, shaimaa hamdy, lecturer of oral periodontology oral medicine and diagnosis, Minia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PVDF membrane in HRA; committee 1059 (Other: ethical committee faculty of dentistry minia university)
Record Dates: First submitted 2025-07-04; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Horizontal Alveolar Bone Loss
Keywords: Horizontal ridge augmentation; PVDF; Titanium Mesh

STUDY DESIGN:
Intervention Model Description: A total of forty-two participants were randomly allocated in a 1:1 ratio into two distinct groups. The control group (n = 21) received a Titanium mesh membrane, which was covered with a collagen membrane, while the study group (n = 21) was treated with a Polyvinylidene fluoride (PVDF) membrane.
  Participants were randomized using a computer-generated method (www.random.org ), ensuring an unbiased distribution of subjects into each group. This process was meticulously overseen by an independent researcher to maintain the integrity of the trial. To further safeguard against bias, allocation concealment was rigorously implemented through the use of sealed, opaque envelopes, which secured the treatment assignments until the point of implementation. This comprehensive approach aimed to enhance the validity and reliability of the research findings.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: PVDF membrane with bone graft used for horizontal ridge augmentation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): This study conducted two main surgical interventions: (T0) one for bone reconstruction and (T1) another for membrane removal following exposure. During the first surgery (T0), patients rinsed with a 0.2% chlorhexidine mouthwash (Eva Pharma, Giza, Egypt) for 60 seconds. All selected sites were anesthetized using articaine hydrochloride 4% with adrenaline (1:100,000) (Artinibsa, Inibsa Spain, Wedjat Pharma). A mid-crestal incision was made, extending to a sulcular incision of adjacent teeth, which included one mesial tooth and two distal teeth. In the edentulous area, the flap extended 3-4 mm posterior to the defect site, along with two vertical releasing incisions. A full-thickness mucoperiosteal flap was raised with a mucoperiosteal elevator (Molt Elevator No. 9, Hu-Friedy®, Hu-Friedy Mfg. Co., LLC. USA) to expose the defect site and adjacent bone; the buccal flap extended apically 5 mm beyond the defect site with a periosteal releasing incision (PRI) for flap mov
  Interventions: Procedure: titanium membrane
- study group (Active Comparator): This study conducted two main surgical interventions: (T0) one for bone reconstruction and (T1) another for membrane removal following exposure. During the first surgery (T0), patients rinsed with a 0.2% chlorhexidine mouthwash (Eva Pharma, Giza, Egypt) for 60 seconds. All selected sites were anesthetized using articaine hydrochloride 4% with adrenaline (1:100,000) (Artinibsa, Inibsa Spain, Wedjat Pharma). A mid-crestal incision was made, extending to a sulcular incision of adjacent teeth, which included one mesial tooth and two distal teeth. In the edentulous area, the flap extended 3-4 mm posterior to the defect site, along with two vertical releasing incisions. A full-thickness mucoperiosteal flap was raised with a mucoperiosteal elevator (Molt Elevator No. 9, Hu-Friedy®, Hu-Friedy Mfg. Co., LLC. USA) to expose the defect site and adjacent bone; the buccal flap extended apically 5 mm beyond the defect site with a periosteal releasing incision (PRI) for flap mov
  Interventions: Procedure: titanium membrane

INTERVENTIONS:
Procedure: titanium membrane — surgical treatment for horizontal ridge augmentation by titanium mesh and PVDF membrane
  Other Names: PVDF membrane; titanium mesh; xenograft bone; collagen membrane

SUMMARY:
This study aims to evaluate the effectiveness of a new PVDF non-resorbable membrane versus Titanium Mesh in the treatment of horizontal ridge defects prepared for implant placement

DETAILED DESCRIPTION:
Alveolar ridge resorption following tooth loss frequently results in horizontal deficiencies that complicate optimal implant placement. To address this, guided bone regeneration (GBR) techniques have become standard in clinical practice, relying on barrier membranes to stabilize graft material and exclude soft tissue interference during healing Titanium mesh membranes have been widely utilized in GBR due to their excellent mechanical strength and ability to maintain space in large or complex defects. Their rigidity ensures stability of the graft material, promoting favorable bone regeneration outcomes. However, the stiffness of titanium meshes can lead to complications such as soft tissue dehiscence and membrane exposure, potentially compromising the regenerative process On the other hand, polyvinylidene fluoride (PVDF) membranes have emerged as a promising alternative in GBR procedures. PVDF is a biocompatible, chemically stable polymer known for its flexibility and resistance to bacterial colonization. Its pliable nature allows for better adaptation to the defect site, potentially reducing the risk of membrane exposure and associated complications. Additionally, the smooth surface of PVDF membranes may minimize soft tissue irritation, further enhancing healing outcomes Materials and methods Study design and patient selection This study was designed as a randomized, controlled, parallel-arm, triple-blinded clinical trial aimed at rigorously comparing the clinical and radiographic outcomes of ridge augmentation procedures utilizing two distinct materials: titanium mesh and high-density polyvinylidene fluoride (PVDF) membrane. In this trial, participants, clinical outcome assessors, and statisticians were kept blind to the treatments being administered to mitigate bias. However, due to the inherent nature of the surgical procedures involved, the operating surgeon could not be blinded.

Participants were selected from the outpatient clinic at the Department of Oral Medicine, Oral Diagnosis, and Periodontology at the Faculty of Dentistry, Nahda University, Beni Suef, Egypt. Inclusion criteria were clearly defined, ensuring that only eligible candidates participated in the study. Prior to enrollment, written informed consent was meticulously obtained from all participants after providing a thorough explanation of the experimental procedures, potential risks, and anticipated benefits associated with their involvement in the research.

The study was conducted in strict adherence to the ethical principles outlined in the Declaration of Helsinki. Additionally, it complied with the International Conference on Harmonization Good Clinical Practice Guidelines. The Research Ethics Committee at the Faculty of Dentistry, Minia University, Minia, Egypt, granted approval for the study, which was registered under a specific registration number ( ) to ensure compliance and transparency in the research process. (clinical trial registration number) 2.2 | Patient Selection

Patient selection underwent stringent selection criteria as follows:

Inclusion criteria:

1. All patients were diagnosed with Class I (Horizontal ridge deficiency) according to Seibert's classification of alveolar ridge deficiencies
2. Maxilla and mandible partial edentulism, not more than 2 teeth missing with D3, D4 bone density

(5) Patients aged 18-55 years. (6) Non-smokers or light smokers (<10 cigarettes/day).

Exclusion Criteria:

(1) Poor oral hygiene with BOP > 20%. (4) Uncontrolled systemic diseases. (5) local and systemic acute infection. (6) Patients who received radiotherapy in the head and neck within the previous five years.

(7) patients with stage III or IV. Randomization and Allocation A total of forty-two participants were randomly allocated in a 1:1 ratio into two distinct groups. The control group (n = 21) received a Titanium mesh membrane, which was covered with a collagen membrane, while the study group (n = 21) was treated with a Polyvinylidene fluoride (PVDF) membrane.

Participants were randomized using a computer-generated method (www.random.org ), ensuring an unbiased distribution of subjects into each group. An independent researcher meticulously oversaw this process to maintain the integrity of the trial. To further safeguard against bias, allocation concealment was rigorously implemented through the use of sealed, opaque envelopes, which secured the treatment assignments until the point of implementation. This comprehensive approach aimed to enhance the validity and reliability of the research findings.

Membrane Preparation Materials: (DMF), using an 80:20 weight ratio of PVDF to PVP. Specifically, 8 grams of PVDF and 2 grams of PVP were added to 90 milliliters of DMF under continuous magnetic stirring at room temperature overnight to ensure complete dissolution and the formation of a uniform solution.

2.6 | Clinical and radiographic assessment All parameters were assessed by the same blinded examiner (A.G) twice: at baseline before surgery (T0) and again after membrane exposure (T1). Data were collected using a specific data collection form.

The primary outcome measured was horizontal bone gain (HBG) (Figure 3a& 6a), determined from a CBCT radiograph taken with the same machine (SCANORA® 3Dx CBCT scanner, Finland). This measurement was evaluated 2 mm below the highest crestal point. At baseline and six months after surgery, the difference between the two measurements was calculated using the formula: HBG (mm) = Postoperative width - Preoperative width.

Secondary outcomes included: the keratinized tissue thickness (KTT), which was measured using an endodontic file No. 8 with a 3 mm diameter silicon stopper. The thickness of the soft tissues was assessed 2 mm apically to the gingival margin. The file was carefully inserted through the soft tissues until a hard surface was felt, keeping it perpendicular to the mucosal surface. Following this, the silicone disk was positioned closely after the file was gently removed from contact with the soft tissue surface, and the penetration depth was then measured (Zucchelli et al., 2013).

Healing complications (HC) were measured, which are classified according to (Fontana et al., 2011) into Class I: No purulent exudate with small membrane exposure (≤ 3 mm), Class II: No purulent exudate with large membrane exposure (> 3 mm), Class III: Both membrane exposure and purulent exudate occur, Class IV: Abscess development without exposure of the membrane. Also, exposure detection could be categorized into early (throughout the first month) or late (after the first month).

Membrane exposure rate (MER): early exposure, before one month (3-29 days), and late exposure, after one month (1-8 months) .

Pseudo-Periosteum Identified (PPI): This parameter was measured at (T1) and classified into Type 1: Typical dense and fibrous, either no tissue or less than 1 mm thick. Type 2: Tissue has moderate consistency and thickness, ranging from 1 to 2 mm. Type 3: Unusual tissue is denser than 2 mm, often vascularized, and has a loose texture Surgical complications (SC) were taken during (T0) A: Inability to close the surgical flaps with the primary intention. B: Flap perforation or laceration. C: Vascular complications: Bleeding after surgery, edema. D: Neurologic complications: Nerve injury during surgery (Fontana et al., 2011).

The flap was closed using a tension-free suture technique that combined horizontal mattress sutures and interrupted sutures, utilizing a 5-0 polypropylene suture (polypropylene monofilament from the industrial zone in Borg El Arab, El Gedida, Alex City, Egypt)

ELIGIBILITY:
Inclusion Criteria:

* All patients were diagnosed with Class I (Horizontal ridge deficiency) according to Seibert's classification of alveolar ridge deficiencies (Seibert, 1983) .Maxilla and mandible partial edentulism, not more than 2 teeth missing with D3, D4 bone density(Smith & Zarb, 1989).
* Presence of a horizontally deficient edentulous ridge (Low < 5 mm) (Misch et al., 2021).
* Good systemic health (ASA I ) (Böhmer et al., 2021).
* Patients aged 18-55 years.
* Non-smokers or light smokers (<10 cigarettes/day).

Exclusion Criteria:

* Poor oral hygiene with BOP > 20%.
* Heavy smoking (more than 10 cigarettes per day).
* local and systemic acute infection.
* Patients who received radiotherapy in the head and neck within the previous five years.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
horizontal ridge augmentation | After 6 months
  determined from a CBCT radiograph taken with the same machine (SCANORA® 3Dx CBCT scanner, Finland). This measurement was evaluated 2 mm below the highest crestal point. At baseline and six months after surgery, the difference between the two measurements was calculated using the formula: HBG (mm) = Postoperative width - Preoperative width.

CONTACTS AND LOCATIONS:
Locations (1):
- Egypt, Cairo, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
After publishing, i will share IPD

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/33380722/